CLINICAL TRIAL: NCT04198480
Title: A Phase I/II, Single Arm, Open Label, Multi-center Clinical Trial to Assess the Efficacy and Safety of JMT103 in Patients With Refractory Hypercalcemia of Malignancy
Brief Title: A Clinical Trial to Assess the Efficacy and Safety of JMT103 in Patients With Refractory HCM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT103CN04
Record Dates: First submitted 2019-11-27; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Hypercalcemia of Malignancy
MeSH Terms: conditions — Humoral Hypercalcemia Of Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JMT103 (Experimental): Eligible subjects will receive JMT103 at a dose of 2 mg/kg subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 2 mg/kg SC on study days 8 and 15.
  Interventions: Drug: JMT103

INTERVENTIONS:
Drug: JMT103 — 2 mg/kg subcutaneously (SC) every 4 weeks with a loading dose of 2 mg/kg SC on study days 8 and 15.

SUMMARY:
The purpose of this study is to determine the potential of JMT103 to treat hypercalcemia of malignancy in patients with elevated serum calcium who do not respond to recent treatment with intravenous bisphosphonates.

DETAILED DESCRIPTION:
This is a Phase I/II, Single arm, Open Label, Multi-center Clinical Trial to Assess the Efficacy and Safety of JMT103 in Patients With refractory Hypercalcemia of Malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed and signed informed consent.
2. Male or female, Adults (>/=18 years).
3. Hypercalcemia of Malignancy (HCM) as defined as documented histologically or cytologically confirmed cancer and a corrected serum calcium (CSC) > 12.5 mg/dL (3.1 mmol /L).
4. Last IV bisphosphonate treatment must be >/= 7 days and </= 30 days before the screening corrected serum calcium; or Last hydration therapy must be >/= 24 hours before the screening corrected serum calcium（Incompatible bisphosphonate）.
5. Adequate organ function.

Exclusion Criteria:

1. Pregnancy.
2. Hyperparathyroidism, or other granulomatous disease.
3. Hepatitis b surface antigen positive.
4. Hepatitis c antibody positive, or HIV antibody positive.
5. Receiving dialysis for renal failure.
6. Known sensitivity to JMT103 composition.
7. Treatment with thiazides, calcitonin, mithramycin, or gallium nitrate within their window of expected therapeutic effect (as determined by the physician) prior to the date of screening CSC.
8. Treatment with cinacalcet within 4 weeks prior to the date of screening CSC.
9. Currently participating another clinical study，or Four weeks or less since receiving an investigational product in another clinical study.
10. In the opinion of the investigator , being unsuitable for inclusion in the study，or subjects withdraw informed consent.
11. Treatment with monoclonal antibody to RANK ligand (RANKL) within 180 days prior to the date of the screening CSC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2020-01-24 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With corrected serum calcium (CSC) ≤ 11.5 mg/dL Within 10 Days after First Dose of JMT103 | 10 Days after First Dose of JMT103
  Percentage of Participants With corrected serum calcium (CSC) ≤ 11.5 mg/dL Within 10 Days after First Dose of JMT103

SECONDARY OUTCOMES:
Percentage of Participants With corrected serum calcium (CSC) ≤ 11.5 mg/dL（2.9 mmol/L） by each visit. | through study completion, an average of 57 Days
  Percentage of Participants With corrected serum calcium (CSC) ≤ 11.5 mg/dL（2.9 mmol/L） by each visit.
Percentage of Participants With corrected serum calcium (CSC) ≤ 10.8 mg/dL（2.7 mmol/L） by each visit. | through study completion, an average of 57 Days
  Percentage of Participants With corrected serum calcium (CSC) ≤ 10.8 mg/dL（2.7 mmol/L） by each visit.
Time to Response | through study completion, an average of 57 Days
  Time to Response
Time to Complete Response | through study completion, an average of 57 Days
  Time to Complete Response
Duration of Response | through study completion, an average of 57 Days
  Duration of Response
Change in Corrected Serum Calcium (CSC) | through study completion, an average of 57 Days
  Change in Corrected Serum Calcium (CSC)
Change in urine N-telopeptide/urine creatinine (uNTx/uCr) | through study completion, an average of 57 Days
  Change in urine N-telopeptide/urine creatinine (uNTx/uCr)

CONTACTS AND LOCATIONS:
Overall Officials: Jin LI, PHD, Principal Investigator — Shanghai East Hospital

IPD SHARING:
Plan to Share IPD: No